CLINICAL TRIAL: NCT03218436
Title: Physical Cold Atmospheric Plasma for the Treatment of Cervical Intraepithelial Neoplasia
Acronym: CAPCIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP CIN
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAP cohort (Active Comparator): Cold Atmospheric plasma intervention
  Interventions: Procedure: CAP treatment
- Control cohort (No Intervention): no intervention

INTERVENTIONS:
Procedure: CAP treatment — Treatment with low-temperature argon plasma during colposcopic examination. No general anesthesia required.
  Arms: CAP cohort

SUMMARY:
Cervical intraepithelial neoplasia will be treated with physical low temperature plasma in the plasma cohort compared to watchful waiting in the control cohort.

Primary endpoint after 3-6 months: Pathological remission.

Secondary endpoint: HPV remission.

DETAILED DESCRIPTION:
The study was completed with Less recruitment as it was planned due to overwhelming study success. The study was published in August 2023. A link has been added to the Reference section.

ELIGIBILITY:
Inclusion Criteria for CAP:

* Histologically confirmed CIN I / II
* Reliable assessment of the radius of the portio and marginal borders of the lesions
* Written consent for treatment with low temperature plasma after reconnaissance

Inclusion Criteria for Control-Group:

* Histologically confirmed CIN I / II
* Reliable assessment of the radius of the portio and marginal borders of the lesions
* Patients who want a waiting procedure and a control examination after 3-6 months

Exclusion Criteria:

* Histologically confirmed CIN III
* Not fully visible transformation zone
* An indication of invasive disease
* Expected lack of compliance of the patient or incapacity of the patient to understand the meaning and purpose of the clinical trial
* Severe cardio-vascular disease
* Lack of patient consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Pathological remission of cervical intraepithelial neoplasia | 3-6 months
  Biopsy, Histopathological examination

SECONDARY OUTCOMES:
Human papilloma virus remission rate | 3-6 months
  Smear testing
Comfort / Dyscomfort during intervention | Immediately, 2 week, 3-6 months
  Freiburger Index of patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Henes, Dr., Principal Investigator — Department for Women's Health; Martin Weiss, Dr., Principal Investigator — Department for Women's Health
Locations (1):
- Department for Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weiss M, Arnholdt M, Hissnauer A, Fischer I, Schonfisch B, Andress J, Gerstner S, Dannehl D, Bosmuller H, Staebler A, Brucker SY, Henes M. Tissue-preserving treatment with non-invasive physical plasma of cervical intraepithelial neoplasia-a prospective controlled clinical trial. Front Med (Lausanne). 2023 Aug 15;10:1242732. doi: 10.3389/fmed.2023.1242732. eCollection 2023. PMID 37654659
- See also: doi: 10.3389/fmed.2023.1242732 — https://pubmed.ncbi.nlm.nih.gov/37654659/